CLINICAL TRIAL: NCT00003634
Title: A Double-Blind Placebo Controlled Trial of Intravenous OvaRex MAb-B43.13 as Post Chemotherapy Consolidation for Ovarian Tubal and Peritoneal Carcinoma
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Residual Disease From Stage III or Stage IV Ovarian Epithelial, Fallopian Tube, or Peritoneal Cancer Following Surgery and Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AltaRex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066718; ALTAREX-OVA-Gy-07; ALTAREX-961452; ALTAREX-OVA-Gy-06; NCI-V98-1488
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — oregovomab

INTERVENTIONS:
Biological: oregovomab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether giving monoclonal antibody therapy is more effective than a placebo in treating patients with ovarian epithelial, fallopian tube, or peritoneal cancer who have responded to surgery and chemotherapy.

PURPOSE: Randomized phase II trial to study the effectiveness of monoclonal antibody therapy in treating patients with residual disease from stage III or stage IV ovarian epithelial, fallopian tube, or peritoneal cancer following surgery and chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the time to disease relapse, survival, and quality of life of patients with stage III or IV ovarian epithelial, tubal, or peritoneal adenocarcinoma treated with OvaRex monoclonal antibody B43.13 OR placebo following complete clinical response to primary therapy. II. Determine the safety of this regimen in these patients. III. Assess the immune response of patients treated with this regimen.

OUTLINE: This is a randomized study. Patients undergo a laparotomy and platinum based chemotherapy prior to randomization. Patients are randomized to 1 of 2 treatment arms: Arm I: Patients receive OvaRex monoclonal antibody B43.13 IV on day 0. Treatment continues at 4, 8, 20, 32, 44, and 56 weeks, and then every 3 months in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive placebo IV on day 0. Placebo administration continues on the same schedule as in arm I. Patients presenting with relapse are provided with second line chemotherapy. Quality of life is assessed at the beginning of the study, after 2 months, and then every 3 months thereafter. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 400 patients (200 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III or IV ovarian epithelial, tubal, or peritoneal adenocarcinoma Must have had complete clinical response to primary therapy consisting of surgical debulking and platinum based chemotherapy Elevated CA 125 (greater than 35 U/mL) prior to or at surgery (if presurgical CA 125 measurement is not available, patient must have a serum CA 125 of at least 100 U/mL and strong tumor tissue expression) Must have residual disease (visible or palpable) at completion of the staging laparotomy (IIIB and IIIC microscopic disease)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 60-100% Life expectancy: At least 6 months Hematopoietic: Hemoglobin at least 8.0 g/dL Lymphocyte count at least 300/mm3 Neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal Renal: Creatinine no greater than 1.6 mg/dL

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 weeks since prior immunotherapy No prior murine monoclonal antibodies for diagnostic or therapeutic purposes Chemotherapy: No more than 1 prior regimen of chemotherapy (change in chemotherapy agents is permitted during primary therapy provided that the change is considered to be part of initial chemotherapy regimen) At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior abdominal, abdominopelvic, or pelvic radiotherapy Surgery: At least 4 weeks since prior surgery No more than 1 interval debulking procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 1998-04

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S. Berek, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (46):
- United States (29):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Wilshire Oncology Medical Center, Pomona, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Patty Berg Cancer Center, Fort Myers, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Saint Mary's Hospital, East Saint Louis, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Alton Ochsner Medical Foundation Hospital, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - North Shore University Hospital, Manhasset, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - University of Texas Southwestern Medical School, Dallas, Texas
  - U.S. Oncology, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Swedish Hospital Tumor Institute, Seattle, Washington
- Canada (17):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Manitoba Cancer Treatment and Research Foundation, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Centre Universitaire de Sante de l'Estrie, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Pavillion de Quebec, Québec, Quebec